CLINICAL TRIAL: NCT03814174
Title: Comparison of Physical Fitness and Activities of the Children With Epilepsy and Their Healthy Peers
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gulsen SIRTBAS, Principal Investigator, Hacettepe University
Other Study IDs: 17/751
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Epilepsy; Physical Activity
Keywords: Childhood Epilepsy; Physical Fitness; Physical Activity; Use of Pedometer
MeSH Terms: conditions — Epilepsy; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate physical fitness and activity levels in children with epilepsy and compare the results with healthy peers.

DETAILED DESCRIPTION:
Many individuals with epilepsy are physically inactive due to the fear of seizures triggered by physical activity/ exercise, and the advices given by the family members and the health care professionals to avoid intense activity . In two studies performed about this subject, this is the probable reason why adult patients with epilepsy have a weaker physical fitness than healthy individuals in the control group. However; in a study of Drawskowski et al., the avoidance of activity and exercise in individuals with epilepsy was investigated, and it was reported that the injuries and seizure problems were rare even during very intense physical activity.

ELIGIBILITY:
Inclusion Criteria:

* children who were diagnosed with epilepsy
* children who can independently continue formal education,
* children who do not need special education
* children who have no additional neurological and neuromuscular disease (epilepsy only)
* children who have a normal or higher cognitive level according to the WISC-R intelligence test
* children who were volunteers to participate in the study
* children whose parents volunteers to participate in the study

Exclusion Criteria:

* The disappearance of volunteerism

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of children with epilepsy and their healthy peers.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Number of steps on pedometer | seven days
  Participants will wear a pedometer (physical activity monitor) for seven consecutive days.
Exercise performance using 6-minute walk test | 1st day (before using device)
  6-minute walk test will be performed in a long, straight, enclosed corridor 30 meters in length. Patients are required to walk in their walking speed with standardized instructions. The distance walked by subjects during 6 minutes will be recorded.
Health-Related Physical Fitness Test for body compozition | 1st day (before using device)
  body mass index
Health-Related Physical Fitness Test for strenght | 1st day (before using device)
  Cadance Based Curl-up Test
Health-Related Physical Fitness Test for balance | 1st day (before using device)
  Flamingo Balance Test
Health-Related Physical Fitness Test for flexibility | 1st day (before using device)
  Sit and Reach Test

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)